CLINICAL TRIAL: NCT04531670
Title: Testing of the Integrated Rapid Access to HIV Prevention Program for People Who Inject Drugs Program
Acronym: iRaPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E20-0596; 1R21DA051934-01A1 (NIH)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: HIV Prevention Program; Opioid-use Disorder
Keywords: People who inject drugs
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iRaPID (Experimental): Participants randomized to the iRaPID program will receive: a) same-day access to PrEP and OAT and educational counseling by the APN; b) safety-check phone calls/SMS; c) follow-up phone call/SMS; and d) clinical visit at Day 30
  Interventions: Behavioral: iRaPID
- Standard of Care (Active Comparator): PWID participants randomized to the training as usual (TAU) will follow the existing clinical guidelines to receive PrEP, OAT, or both.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: iRaPID — Participants randomized to the iRaPID program will receive: a) same-day access to PrEP and OAT and educational counseling by the APN; b) safety-check phone calls/SMS; c) follow-up phone call/SMS; and d) clinical visit at Day 30
  Arms: iRaPID
Other: Standard of Care — PWID participants randomized to the training as usual (TAU) will follow the existing clinical guidelines to receive PrEP, OAT, or both.
  Arms: Standard of Care

SUMMARY:
This is a pilot study of an integrated rapid access HIV prevention program for People who inject drugs (PWID) called iRaPID. The program incorporates same-day access to Pre-exposure Prophylaxis (PrEP) and Opioid Agonist Therapy (OAT).

DETAILED DESCRIPTION:
A Hybrid type 1 implementation science design,will be used to pilot test the APN-led iRaPID program while exploring information on its implementation at multiple time points through the study. The hybrid type 1 pilot trial provides an implementation heuristic to assess potential research questions, perhaps more comprehensively, accurately and certainly earlier than could be achieved in a sequential 'intervention-then-preliminary-pilot study' strategy. In this hybrid type 1 pilot trial, the RCT will be utilized to:

* Examine feasibility and acceptability among PWID and clinical stakeholders for an adapted APN-delivered, rapid HIV prevention program for PWID (iRaPID) that integrates same-day PrEP and OAT.
* Estimate the preliminary efficacy of PrEP and OAT uptake in a pilot randomized controlled trial of the iRaPID vs. treatment as usual strategy in PWID without HIV.

To assess future scale-up factors, the Consolidated Framework for Implementation Research (CFIR) will be utilized with the nominal group technique (NGT). It is a conceptual framework developed to guide the assessment of multilevel implementation contexts. The CFIR framework was selected because it provides a structured menu of constructs associated with effective implementation. It consists of 5 domains with 39 underlying constructs. As recommended by Damschroder, in this study 8 CFIR constructs based on the relevancy will be measured.

During the NGT, participants will be asked questions related to the multi-level implementation factors that will be based on the sample guide available on http://cfirguide.org but tailored for PWID. After posing each question, participants silently generate individual ideas. Then, using a round-robin elicitation process, each person contributes ideas that are recorded visually. They then engage in group discussion to clarify and evaluate the ideas. Items are then grouped by consensus with duplicate items removed. Then, each participant casts three votes on items as they deem them important. Votes are immediately tallied, ranked based on total number of votes, and the facilitator leads a final discussion to review the results. Sessions will take 60 minutes and be audio-recorded and transcribed.

ELIGIBILITY:
Inclusion Criteria:

PWID

1. Age ≥18 years
2. HIV-negative
3. Reporting injection drug use (past 3 months)
4. Substantial ongoing risk for HIV acquisition
5. OUD based on the DSM-V criteria

Stakeholders

1. Age ≥18 years
2. APNs, patient navigators, counselors, and administrators who reflect the range of characteristics of staff members that are involved in HIV care to PWID

Exclusion Criteria:

PWID and stakeholders

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unable to provide informed consent
2. Unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility - participants screened | 6 months
  The number of participants screened will be used as a measure of feasibility
Feasibility - participants recruited | 6 months
  The number of participants recruited will be used as a measurement of feasibility
Feasibility - participants randomized | 6 months
  The number of participants randomized will be used as a measurement of feasibility
Feasibility - participants retained | 6 months
  The number of participants retained will be used as a measurement of feasibility
Feasibility - treatment adherence | 6 months
  The number of participants that adhere to treatment will be used as a measurement of feasibility
Acceptability | 6 months
  Acceptability will be measured using a 10-item acceptability rating profile. Acceptability will be based on descriptive statistics from the acceptability measures (score ≥70) and analysis of qualitative data, which will be done using thematic analysis
Uptake of PrEP and OAT | 6 month
  PrEP uptake proportion at 6-month follow-up will be estimated and compared using linear contrast statement in SAS.
Adherence to PrEP | 6 months
  Adherence to PrEP will be measured using the visual analogue scale and dried blood spots
Persistence on PrEP | 6 months
  Persistence on PrEP will be measured by collecting information on refilled within 30 days after exhausting PrEP from previous fill data

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Clinical and Community Research, New Haven, Connecticut, United States

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Derived] Khati A, Altice FL, Vlahov D, Eger WH, Lee J, Bohonnon T, Wickersham JA, Maviglia F, Copenhaver N, Shrestha R. Nurse Practitioner-Led Integrated Rapid Access to HIV Prevention for People Who Inject Drugs (iRaPID): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 11;11(10):e42585. doi: 10.2196/42585. PMID 36222826